CLINICAL TRIAL: NCT00708942
Title: A Randomized Phase II Study of Hexaminolevulinate (HAL) Photodynamic Therapy (PDT) in Patients With Low-grade Cervical Intraepithelial Neoplasia (CIN1)
Brief Title: Hexaminolevulinate (HAL) Photodynamic Therapy (PDT) of Cervical Intraepithelial Neoplasia (CIN) Grade 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment, study stopped with only 13 of 70 patients included in second part of the study
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC CE201/08
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2013-04-15 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical intraepithelial neoplasia (CIN)
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator): HAL suppository (single administration, HAL 100mg), laser illumination (50J/cm2)
  Interventions: Drug: Hexaminolevulinate (HAL)
- 2 (Placebo Comparator): Placebo suppository (single administration), laser illumination (50J/cm2)
  Interventions: Drug: Placebo
- 3 (No Intervention)
- 4 (Active Comparator): HAL ointment (5%, 100mg, single administration), LED diode illumination (50J/cm2)
  Interventions: Drug: Hexaminolevulinate (HAL)
- 5 (Placebo Comparator): Placebo ointment (single administration), no illumination
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hexaminolevulinate (HAL) — Drug: hexaminolevulinate (HAL) Suppository HAL 100 mg for 3-7 hours application
  Arms: 1
Drug: Placebo — Placebo suppository, for 3-7 hours application
  Arms: 2
Drug: Hexaminolevulinate (HAL) — Drug: hexaminolevulinate (HAL) Ointment HAL 100 mg for 5 hours application
  Arms: 4
Drug: Placebo — Placebo ointment for 5 hours application
  Arms: 5

SUMMARY:
The study will examine the effect of HAL vs placebo photodynamic therapy of low-grade cervical precancerous lesions (dysplasia) in women.

DETAILED DESCRIPTION:
Low-grade cervical intraepithelial neoplasia (CIN1) is caused by persistent HPV infection and may worse case develop into cancer. In most cases both the virus infection and lesions (CIN1) regress spontaneously, but must be followed up with gynecological examinations to ensure normalization. If further persistent disease and worsening to precancerous lesions (CIN2-3), the usual treatment is surgery, where one removes the tissue in the cervix where the CIN lesions are.

In this research study we will evaluate a new non-surgical treatment for CIN1 using hexaminolevulinate (HAL) photodynamic therapy (PDT). HAL PDT is the combination of a medication and a specific type of light to activate the drug. HAL PDT selectively removes CIN lesions while preserving normal tissue, thus this may be an alternative to frequent gynecological consultations and local surgery that may have undesirable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Satisfactory colposcopy examination
* Negative endocervical canal by colposcopy
* Ectocervical CIN1 as verified by local pathologist (biopsy).
* Colposcopical visible lesion at visit 2, before photoactivation
* Written Informed Consent signed
* Age 18 or above

Exclusion Criteria:

* Previous treatment of CIN or invasive disease or suspicion of either micro-invasive or invasive disease
* Malignant cells on cytology or histology
* Atypical glandular cells (AGC) or adenocarcinoma in situ (AIS) on cytology
* Suspicion of endocervical disease on colposcopy
* Current pelvic inflammatory disease, cervicitis, or other gynecological infection as per colposcopy and clinical examination
* Known or suspected porphyria
* Known allergy to hexaminolevulinate or similar compounds (e.g. methyl aminolevulinate or aminolevulinic acid)
* Use of heart pacemaker
* Pregnancy
* Nursing
* Childbirth or miscarriage within six weeks of enrolment - Known
* Participation in other "competitive" clinical studies either concurrently or within the last 30 days
* Risk of poor protocol compliance
* Not willing to use adequate birth control from screening until last PDT
* Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hillemanns, MD, PhD, Principal Investigator — Medizinische Hochschule Hannover, Hannover, Germany
Locations (5):
- Department of Obstetrics and Gyneacology, Lille University Hospital, Lille, France
- Department of Obstetrics and Gynecology, Hanover, Germany
- Norway (3):
  - Fritzøe klinikk, Larvik
  - Department of Obstetrics and Gynaecology, Ullevål University Hospital, Oslo
  - Medicus, Trondheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects recruited from medical clinics/hospitals. Start of recruitment arms 1-3: Jan 2009 End of recruitment arms 1-3: Feb 2010 Start of recruitment arms 4-5: Nov 2010 End of recruitment arms 4-5: Jul 2011
Pre-assignment Details: Recruitment to part 1, including arms 1-3, completed before initiation of part 2 (arms 4-5). Arms 4 and 5 was a protocol amendment.
Period: Overall Study
Arm/Group | Arm 1: HAL Suppository, Laser Illumination | Arm 2: Placebo Suppository, Laser Illumination | Arm 3: No Intervention | Arm 4: HAL Ointment, LED Diode Illumination | Arm 5: Placebo Ointment, no Illumination
Started | 47 | 12 | 11 | 10 | 3
Completed | 40 | 11 | 9 | 10 | 2
Not Completed | 7 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: HAL Suppository, Laser Illumination | Arm 2: Placebo Suppository, Laser Illumination | Arm 3: No Intervention | Arm 4: HAL Ointment, LED Diode Illumination | Arm 5: Placebo Ointment, no Illumination | Total
Number analyzed (Participants) | 47 | 12 | 11 | 10 | 3 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 47 | 12 | 11 | 10 | 3 | 83
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 30.2 (6.9) | 29.1 (4.7) | 32.5 (8.4) | 38.8 (9.4) | 31.0 (4.0) | 31.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 12 | 11 | 10 | 3 | 83
  Male | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 7 | 1 | 1 | 1 | 0 | 10
  Norway | 0 | 1 | 0 | 9 | 3 | 13
  Germany | 40 | 10 | 10 | 0 | 0 | 60

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Based on histology, cytology and HPV status. "Complete response" is defined as normal pathology, normal cytology and negative HPV.
Time Frame: 6 month
Population: Per protocol population. Patients with major protocol violations excluded.
Measure: Number; unit: percentage of no. of patients analyzed
Arm/Group | Arm 1: HAL Suppository, Laser Illumination | Arm 2: Placebo Suppository, Laser Illumination | Arm 3: No Intervention | Arm 4: HAL Ointment, LED Diode Illumination | Arm 5: Placebo Ointment, no Illumination
Number analyzed (Participants) | 35 | 10 | 6 | 10 | 3
percentage of no. of patients analyzed | 57.1 (0) | 40.0 (0) | 0.0 (0) | 90.0 (0) | 33.3 (0)

2. Secondary Outcome: Eradication of HPV
Description: High risk HPV
Time Frame: 6 months
Population: Patients who were positive for high risk HPV at baseline
Measure: Number; unit: percentage of no. of patients analyzed
Arm/Group | Arm 1: HAL Suppository, Laser Illumination | Arm 2: Placebo Suppository, Laser Illumination | Arm 3: No Intervention | Arm 4: HAL Ointment, LED Diode Illumination | Arm 5: Placebo Ointment, no Illumination
Number analyzed (Participants) | 20 | 7 | 3 | 4 | 3
percentage of no. of patients analyzed | 60.0 (0) | 28.6 (0) | 100 (0) | 50.0 (0) | 33.3 (0)

3. Secondary Outcome: Incidence of Patients With Adverse Events
Time Frame: 3 months
Population: All patients treated
Measure: Number; unit: percentage of no of patients analyzed
Arm/Group | Arm 1: HAL Suppository, Laser Illumination | Arm 2: Placebo Suppository, Laser Illumination | Arm 3: No Intervention | Arm 4: HAL Ointment, LED Diode Illumination | Arm 5: Placebo Ointment, no Illumination
Number analyzed (Participants) | 47 | 12 | 11 | 10 | 3
percentage of no of patients analyzed | 44.7 | 25.0 | 18.2 | 70.0 | 66.7

ADVERSE EVENTS:
Arm/Group | Arm 1: HAL Suppository, Laser Illumination | Arm 2: Placebo Suppository, Laser Illumination | Arm 3: No Intervention | Arm 4: HAL Ointment, LED Diode Illumination | Arm 5: Placebo Ointment, no Illumination
Serious Adverse Events (participants affected / at risk) | 3/47 | 0/12 | 1/11 | 0/10 | 0/3
Other Adverse Events (participants affected / at risk) | 16/47 | 3/12 | 1/11 | 6/10 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: HAL Suppository, Laser Illumination (N=47) | Arm 2: Placebo Suppository, Laser Illumination (N=12) | Arm 3: No Intervention (N=11) | Arm 4: HAL Ointment, LED Diode Illumination (N=10) | Arm 5: Placebo Ointment, no Illumination (N=3)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concomitant disease aggravated (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: HAL Suppository, Laser Illumination (N=47) | Arm 2: Placebo Suppository, Laser Illumination (N=12) | Arm 3: No Intervention (N=11) | Arm 4: HAL Ointment, LED Diode Illumination (N=10) | Arm 5: Placebo Ointment, no Illumination (N=3)
Uterine pain (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Slow recruitment lead to early terminaiton of the second part of the trial, including arms 4 and 5, after enrolment of 13 patients. No formal statistical analysis conducted on this part of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may publish the results from his/her site, provided that the publication does not disclose confidential information or interfere with sponsor's efforts to obtain patent protection for inventions. The sponsor must receive material for review not less than sixty (60) days prior to their proposed submission.

In this multi center study, collective publications are anticipated. The PI must not independently publish the results of the Study before the first collective publication.